CLINICAL TRIAL: NCT04009512
Title: Visceral Manifold Study for the Repair of Thoracoabdominal Aortic Aneurysms
Brief Title: Endovascular Repair of Thoracoabdominal Aortic Aneurysms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Eagleton (Other)
Collaborators: Medtronic (Industry); NAMSA (Other); Sanford Health (Other)
Responsible Party: Sponsor-Investigator, Matthew Eagleton, Chief, Division of Vascular and Endovascular Surgery, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-01-001
Record Dates: First submitted 2019-06-24; First posted 2019-07-05 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Thoracoabdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Primary Study Arm (Experimental): The Valiant Thoracoabdominal Stent Graft System is comprised of two investigational devices including the Thoracic Bifurcate and the Visceral Manifold. These devices work to facilitate endovascular stenting of the visceral vessels (renals, celiac, SMA) while maintaining flow to the visceral and infrarenal segments.
  Interventions: Device: Valiant Thoracoabdominal Stent Graft System
- Expanded Use Arm (Experimental): The Valiant Thoracoabdominal Stent Graft System is comprised of two investigational devices including the Thoracic Bifurcate and the Visceral Manifold. These devices work to facilitate endovascular stenting of the visceral vessels (renals, celiac, SMA) while maintaining flow to the visceral and infrarenal segments. The expanded use arm provides broaden inclusion criteria to include select patients excluded from the primary study arm.
  Interventions: Device: Valiant Thoracoabdominal Stent Graft System

INTERVENTIONS:
Device: Valiant Thoracoabdominal Stent Graft System — This system of devices works to facilitate endovascular stenting of the visceral vessels (renals, celiac, SMA) while maintaining flow to the visceral and infrarenal segments in patients with thoracoabdominal aneurysms.

SUMMARY:
The primary objective of this study is to assess the use of the thoracic bifurcation and the visceral manifold devices in the repair thoracoabdominal aortic aneurysms in patients with appropriate anatomy. The primary intent of the study is to assess safety and preliminary effectiveness of the device. Additionally, the study will assess technical success and treatment success at each follow-up interval.

DETAILED DESCRIPTION:
The primary objective is to assess the use of the thoracic bifurcation and the visceral manifold stent graft system to repair thoracoabdominal aortic aneurysms in patients with appropriate anatomy. The primary intent of the study is to assess safety (i.e. freedom from major adverse events (MAE) at 30 days) and preliminary effectiveness (i.e., treatment success and technical success) of the device (i.e., the proportion of treatment group subjects that achieve and maintain treatment success at one year). Additionally, the study will assess technical success and treatment success at each follow-up interval.

ELIGIBILITY:
Inclusion Criteria:

Primary Arm Inclusion Criteria:

A patient may be entered into the study if the patient has at least one of the following:

* An aneurysm with a maximum diameter of > 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
* Aneurysm with a history of growth > 0.5 cm in 6 months
* Saccular aneurysm deemed at significant risk for rupture
* Symptomatic aneurysm greater than or equal to 4.5 cm

Other inclusion criteria

* Axillary or brachial and iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
* Proximal landing zone for the thoracic bifurcation stent graft that has:

  * ≥ 2.5 cm of nonaneurysmal aortic segment including previously placed graft material (neck) distal to the left subclavian artery (LSA) and a diameter in the range of 26-42 mm
  * Adequate distance from the celiac artery, in order to accommodate cannulation from the antegrade access point when considering the total deployed length of the thoracic bifurcation and visceral manifold
* Iliac artery or aortic distal fixation site, including both native tissue and previously placed graft, greater than or equal to 15 mm in length and diameter in the range of 8 - 25 mm
* Age: ≥ 18 years old
* Life expectancy: > 1 year

Exclusion Criteria:

Primary Arm Exclusion criteria

* Patient is a good candidate for and elects for open surgical repair
* Can be treated in accordance with the instructions for use with a legally marketed endovascular prosthesis
* Is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent by patient or legal representative
* Urgent or emergent presentation
* Patient is pregnant or breastfeeding
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a dissection in the portion of the aorta intended to be treated
* Obstructive stenting of any or all of the visceral vessels
* Poor performance status including two major system failures (including but not limited to cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)

Medical exclusion criteria

* Known sensitivities or allergies to the materials of construction of the devices, including nitinol (Nickel: Titanium), polyester, platinum-iridium, polytetrafluoroethylene (PTFE), platinum, gold, polyethylene, or stainless steel.
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
* Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection
* Baseline creatinine greater than or equal to 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome)
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in a landing zone that expands beyond any limits of the previously placed graft material

Anatomical exclusion criteria

* Minimum branch vessel diameter less than 5 mm
* Thrombus or excessive calcification within the proximal aortic neck
* Anatomy that would not allow maintenance of at least one patent hypogastric artery
* Anatomy that would not allow primary or assisted patency of the left subclavian artery

Expanded Use Arm Inclusion Criteria

Patient that meet the criteria for inclusion in the primary study arm but has one or more of the following criteria which would exclude them from the primary study arm:

An expanded use arm of the study will broaden inclusion criteria to include patients with the following :

* Minimum branch vessel diameter <5mm
* Urgent or emergent presentation
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a type B dissection (subacute or chronic) in the portion of the aorta intended to be treated
* Poor performance status including two major system failures (including but not limited to cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)
* Baseline creatinine greater than or equal to 2.0 mg/dL
* Anatomy that does not allow maintenance of at least one hypogastric artery
* Anatomy that does not allow primary or assisted patency of the left subclavian artery
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in a landing zone that expands beyond any limits of the previously placed graft material
* Obstructive stenting of any or all of the visceral vessels
* Patient that meets the criteria for inclusion in the primary study arm and:

  * Would not be eligible for the primary study arm per a documented reason other than those outlined above, and
  * Per the opinion of the Principal Investigator, with concurrence of the IRB, alternative therapies are unsatisfactory and the probable risk of using the investigational device is no greater than the probable risk from the disease or condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2026-08-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Freedom from MAEs (at 30 Days) | 30 Days post- procedure
  Major Adverse Events include: all-cause mortality within 30 days of the procedure, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and stroke.
Preliminary Effectiveness (treatment and technical success) | 1- year post-procedure
  Treatment success is defined as a composite of technical success and freedom from the following:
  * Aneurysm enlargement i.e., >5mm as compared to any previous CT measure using orthogonal (i.e., perpendicular to the centerline) measurements
  * Aneurysm rupture
  * Aneurysm-related mortality
  * Conversion to open repair
  * Secondary intervention for migration, Type I and III endoleaks, device integrity failure (e.g., fracture), and patency-related events (i.e., device component stenosis or occlusion and embolic events)

SECONDARY OUTCOMES:
Technical Success | at each follow-up interval (five years)
  Technical success and the individual components of technical success include:
  * Successful delivery
  * Deployment at the intended implantation site
  * Patency of all endovascular graft and stent components
  * Absence of device deformations requiring unplanned placement of an additional device
  * Absence of inadvertent covering of aortic branch vessels
  * Successful withdrawal
Treatment Success | at each follow-up interval (five years)
  Treatment success and the individual components of treatment success including freedom from the following at each follow-up interval:
  * Aneurysm enlargement
  * Aneurysm-related mortality
  * Aneurysm rupture
  * Conversion to open repair
  * Secondary intervention for migration, type I and III endoleaks, device integrity failure (i.e., fracture), and patency-related events (i.e., device stenosis or occlusion and embolic events).
  * Renal failure
  * All-cause mortality
  * Endoleaks
  * Device integrity failure (e.g., fracture)
  * Patency-related events (i.e., device stenosis or occlusion and embolic events)
  * Other device-related events

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States